CLINICAL TRIAL: NCT00162851
Title: A Pilot Study to Evaluate the Safety of Subcutaneous Alemtuzumab (MabCampath, Campath) in Patients With B-Cell Chronic Lymphocytic Leukemia
Brief Title: Study to Evaluate the Safety of Subcutaneous Alemtuzumab in Patients With B-Cell Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Schering Nordiska AB (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM219
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2005-08

CONDITIONS: B-CLL
MeSH Terms: interventions — Alemtuzumab

INTERVENTIONS:
Drug: alemtuzumab

SUMMARY:
This is a Phase II trial to study the safety and tolerability of subcutaneous alemtuzumab administered without dose escalation to patients with advanced B-cell chronic lymphocytic leukemia (B-CLL).

ELIGIBILITY:
Inclusion Criteria:

* B-CLL that has failed fludarabine

Exclusion Criteria:

* Performance status grade 3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-04; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders C Osterborg, Professor, Principal Investigator — Dept. of Hematology, Karolinska University Hospital
Locations (1):
- Dept. of Hematology, Karolinska University Hospital, Stockholm, Sweden